CLINICAL TRIAL: NCT04846075
Title: The Effect of Ramadan on the Blood Concentration of Serotonin, Dopamine, Brain-Derived Neurotorophic Factor and Nerve Growth Factor: A Replication Study
Brief Title: Biological and Psychological Health Effect of Ramadan Study
Acronym: HERS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bastyr University (Other)
Responsible Party: Principal Investigator, Masa Sasagawa, ND, PhD, Assistant Research Scientist, Bastyr University
Other Study IDs: 21-1690
Record Dates: First submitted 2021-04-08; First posted 2021-04-15 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Quality of Life
MeSH Terms: interventions — phosphoribosylanthranilate isomerase; Social Work; Poverty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 10 mL serum (SST) and 10 mL (plasma) EDTA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ramadan Group: Diurnal fasting and spiritual practices. Operationally assessed by the level of compliance to Sawm, Salat, and Zakat.
  Interventions: Behavioral: Ramadan fasting, praying, and welfare for poor

INTERVENTIONS:
Behavioral: Ramadan fasting, praying, and welfare for poor — Abstaining from food, drink, smoking, and sexual activity duirng daytime; ritualistic praying at specific time of a day for five or more times; volunteering for communities or donation
  Other Names: Diurnal fasting or Sawm; five or more prayers or Salat; donation or volunteering or Zakat

SUMMARY:
This observational study collects data on blood neurotransmitter and neuromodulator levels of subjects observing Ramadan. Additional information collected are a diet record, mood and perceived stress using validated surveys at three time points: a) before starting Ramadan, b) at the midpoint evaluation, and c) at the end of Ramadan. Three additional dispositional factors collected at the beginning and at the end are: a) sense of belonging, b) purpose in life (sense of coherence), and c) empathy (interpersonal reactivity index). The subjects are also individually interviewed on their experience of Ramadan as narrative data.

DETAILED DESCRIPTION:
This is an observational study seeking research volunteers during Ramadan in the Pacific Northwest. We plan to recruit 10 female and 5 male volunteers. Each subject will donate her/his blood (20 milliliters) at three time points: a) before initiation of Ramadan, b) 14 days later, and c) 30 days later (60 milliliters total over one month). Because the dates of Ramadan in 2021 occur on April 12th through May 11th, the three days of the blood collection will be April 10th, April 27th and May 11th ± 1 day. Due to current COVID-19 restrictions, mass gatherings at mosque do not happen. This study deploys a mobile phlebotomist who is a licensed healthcare practitioner who will set up a droplet barrier phlebotomy station. The time of phlebotomy is determined based on the hydration status of each individual. The specimens will be packed in an ice cooler and processed (centrifuged and divided into aliquots) at Bastyr University Tierney laboratory and stored in a -80 degree Celsius freezer until analyzed at the same time for the three time points. Narrative data will also be collected through individual conversations (phone or in-person) at the completion of Ramadan, reflecting on the study and any heightened sense of spirituality.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age at the time of baseline blood draw, up to 65 years old
* Community member who observe Ramadan during April 12 (Monday evening) through May 11, 2021 (Tuesday sundown)
* Understand and sign the informed consent form and have ability to comply with the requiremnets of the study
* Vaccinated for COVID or having a history of a positive PCR test which was resolved

Exclusion Criteria:

* Anticubital vein is not accessible
* Pregnant, breastfeeding, recovering from major illness or surgery that influences quality of life
* Who reside more than 14 miles away from the city limits
* Unavailable to meet in-person and donate blood for any of three measurement days (basline, 15th day, post Ramadan)
* Smoking, drinking aclohol or using recreational drug
* Presence of a condition that in the opinon of the Investigator would compromise the safety of the participant or the quality of the data

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Upon obtaining permission from the community leaders (Muslim Association of Puget Sound) and support from IMAN Center of Kirkland, flyers will be disseminated through friends and family members of Muslim members. Anyone who observes Ramadan for religious or health reasons, and who are also committed to following the fasting as prescribed, and who do not have chronic health conditions, will be eligible for participation in this study.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2021-04-08 (Actual); Primary Completion 2021-05-15 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in dopamine concentration | 0 to 30 days
  Plasma dopamine level pg/mL
Change in serotonin concentration | 0 to 30 days
  Plasma serotonin level ng/mL
Change in Brain-Derived Neurotrophic factor (BDNF) concentration | 0 to 30 days
  Plasma BDNF level pg/mL
Change in Nerve Growth Factor (NGF) concentration | 0 to 30 days
  Plasma NGF level pg/mL

SECONDARY OUTCOMES:
Change in mood measured by Positive And Negative Affect Scale (PANAS) | 0 to 30 days
  PANAS questionnaire in English
Change in perceived stress level measured by Weekly Stress Inventory (WSI) | 0 to 30 days
  Weekly Stress Inventory in English

CONTACTS AND LOCATIONS:
Overall Officials: Masa Sasagawa, ND, PhD, Principal Investigator — Bastyr University
Locations (1):
- Bastyr University, Kenmore, Washington, United States

IPD SHARING:
Plan to Share IPD: No
Data are collected by subject IDs (SIDs). Only aggregate results will be available